CLINICAL TRIAL: NCT03320408
Title: Predicting Aneurysm Growth and Rupture With Longitudinal Biomarkers (PARIS Study) & Biobank Pearl AAA
Brief Title: Predicting Aneurysm Growth and Rupture With Longitudinal Biomarkers
Acronym: PARIS
Status: Completed | Type: Observational
Sponsor: Ron Balm (Other)
Responsible Party: Sponsor-Investigator, Ron Balm, Principal Investigator, Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Organization: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Other Study IDs: NL59991.018.17; Biobank Pearl AAA (Registry Identifier: Biobank Pearl AAA)
Record Dates: First submitted 2017-10-12; First posted 2017-10-25 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Abdominal Aortic Aneurysm; Abdominal Aortic Aneurysm, Ruptured
Keywords: biobank; pathogenesis; Aortic Aneurysm
MeSH Terms: conditions — Aortic Aneurysm, Abdominal; Rupture; Aortic Aneurysm

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 10 Years
Biospecimen Retention: Samples With DNA — Three types of biospecimens will be collected, depending on the clincial stage of the abdominal aortic aneurysm.
  Blood:
  EDTA plasma; Serum; Citrate plasma; EDTA for DNA; PAXgene for RNA.
  Urine.
  Aneurysm tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Asymptomatic AAA: These patients will be included while their AAA is asymptomatic and while they are under surveillance by their vascular surgeon.
- Acute AAA: These are the patients that are included while they presented in the participating hospitals because either a symptomatic or ruptured AAA. For this group, a different recruitment procedure exists which has been approved by the appropriate medical ethical committee.
- Repaired AAA: These patients are included while they already had had AAA repair (both elective and emergency repair).

SUMMARY:
First aim: PARIS study

The main aim of the current study is to determine the association between abdominal aortic aneurysm (AAA) progression and the evolution of proteases and cytokines levels.To achieve this aim, we will prospectively collect blood, aortic tissue, patient data, and imaging data. Aortic tissue will only be obtained when patients undergo conventional open repair. The other biomaterials will be collected during regular patient follow-up visits, with a maximum frequency of once per year.

Second aim: Pearl AAA biobank

For future research purposes, a new biobanking infrastructure will be created to collect and store additional blood and urine samples in a biobank. This biobank will be embedded within the infrastructure of the 'Parelsnoer Institute' (PSI) and will be called Pearl AAA. The Pearl AAA will be established in the extension of the PARIS study

DETAILED DESCRIPTION:
The PARIS study aims to determine the correlation between AAA progression (growth or rupture) and the evolution of serum levels of proteases and cytokines over time. A repeated measures analysis will be done to use all longitudinal data available.

The Pearl AAA biobank will be established to enable the PARIS study, but also aims to facilitate future research. Such future research should fall under the scientific aims of the Pearl AAA, which are:

* To gain insight in the pathogenesis of AAA
* To gain more knowledge in the rupture risk of AAA
* To evaluate and potentially improve treatment of AAA

The 'Parelsnoer Institute' will facilitate the biobank Pearl AAA with certain aspects such as, but not limited to the following:

* Standardized operating procedures for the collection and storage of the biosamples across all participating hospitals
* Information architect to establish a data dictionary in which all variables are defined
* Standardized procedures for coding of patient data before storage
* Standardized digital infrastructure to enhance storage of patient data and imaging data

ELIGIBILITY:
Inclusion Criteria:

* Adult participant (18 years or older)
* Participant has an AAA or has previously been treated for an AAA
* Adequate comprehension of the Dutch language to provide written informed consent

Exclusion Criteria:

* A patient who is decisionally impaired. The only exception to this are the patients who are decisionally impaired due to the effects of an acute AAA. This particular group is eligible for which a separate recruitment and consent procedure exists.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients with an abdominal aortic aneurysm who present themselves in the participating hospitals.
Sampling Method: Probability Sample
Enrollment: 790 (Actual)
Dates: Start 2017-10-04 (Actual); Primary Completion 2023-08-04 (Actual); Study Completion 2023-08-04 (Actual)

PRIMARY OUTCOMES:
AAA growth | Up to 10 years of follow-up
  Growth of abdominal aortic aneurysm, measured on imaging made for clinical purposes
AAA rupture | Up to 10 years of follow-up
  Rupture of an abdominal aortic aneurysm
Death | Up to 10 years of follow-up
  All-cause mortality
Evolution of serum levels of proteases | a maximum of 1 measurement annually up to 10 years of follow-up
  Repeated measurements analysis of serum levels of proteases in cohort of asymptomatic AAAs
Evolution of serum levels of cytokines | a maximum of 1 measurement annually up to 10 years of follow-up
  Repeated measurements analysis of serum levels of cytokines in cohort of asymptomatic AAAs
Protease levels in aortic tissue | If open AAA repair is performed and aortic tissue is collected, protease levels will then be measured. This is a one-time measurement.
  Protease levels in aortic tissue
Cytokine levels in aortic tissue | If open AAA repair is performed and aortic tissue is collected, cytokine levels will then be measured. This is a one-time measurement.
  Cytokine levels in aortic tissue

SECONDARY OUTCOMES:
Type of complications after AAA repair | Will be measured up to 10 years after AAA repair is performed
  Type of complications using methodology from the Dutch committee of the "Nederlandse Vereniging voor Heelkunde," named the "Landelijke Heelkunde Complicatie Registratie" as found on www.lhcr.nl
Incidence of complications after AAA repair | Will be measured up to 10 years after AAA repair is performed
  Number of complications after abdominal aortic aneurysm repair

CONTACTS AND LOCATIONS:
Overall Officials: Ron Balm, MD PhD, Principal Investigator — Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Locations (2):
- Netherlands (2):
  - Leiden University Medical Center (LUMC), Leiden, South Holland
  - Department of Vascular Surgery, Amsterdam UMC, location AMC, Amsterdam

IPD SHARING:
Plan to Share IPD: Yes
Researchers can initiate the procedure to request IPD for research that falls within the scientific scope of the biobank Pearl AAA.
Time Frame: Depending on the specific study protocols that are submitted to the biobank Pearl AAA
Access Criteria: Procedural criteria can be attained by contacting the researchers.

REFERENCES:
- [Derived] Jalalzadeh H, Indrakusuma R, Blankensteijn JD, Wisselink W, Yeung KK, Lindeman JHN, Hamming JF, Koelemay MJW, Legemate DA, Balm R. Design and protocol of a comprehensive multicentre biobank for abdominal aortic aneurysms. BMJ Open. 2019 Aug 1;9(8):e028858. doi: 10.1136/bmjopen-2018-028858. PMID 31375618